CLINICAL TRIAL: NCT03542604
Title: The Effects of Treating Insomnia Prior to a Weight Loss Intervention in Women With Early Stage Breast Cancer
Brief Title: Cancer, Obesity/Overweight and Insomnia Study
Acronym: COIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Under Armour, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: J17120; IRB00132883 (Other: JHU IRB)
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer; Overweight and Obesity; Insomnia
MeSH Terms: conditions — Breast Neoplasms; Overweight; Obesity; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: A total of 30 participants will be randomized to either cognitive-behavioral treatment for insomnia with behavioral weight loss (CBT-I+BWL) or a sleep education control condition with behavioral weight loss (EDU+BWL). The EDU group will have study sessions spread out in a similar fashion to the CBT-I group, and clinical outcomes will be compared between groups at baseline, 8 weeks (after the CBT-I or EDU program) and at 3 and 6 months after starting BWL. The primary outcome will be % total weight loss. Additionally, eating behaviors, physical activity, and sleep parameters will be carefully assessed.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Participants will not be blinded to the intervention assignment. However, data collection of anthropometric measurements (including height, weight, hip and waist circumference) will be done by a study member blinded to the randomization. Since participants will be aware of their intervention assignment, there are no anticipated circumstances for breaking the blinding or planned procedures for breaking the blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I + BWL (Experimental): Cognitive behavioral therapy intervention for insomnia: 6 sessions over 8-week period combining education and behavioral techniques to reduce insomnia. Sleep intervention followed by behavioral weight loss intervention.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- EDU + BWL (Placebo Comparator): Program will parallel the CBT-I intervention in number and length of sessions. Intended to disseminate basic information about sleep, including behavioral treatment information that is widely available to patients and practitioners.Will be followed by behavioral weight loss intervention.
  Interventions: Behavioral: Sleep Education

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — CBT-I involves identifying and replacing thoughts and behaviors that cause or worsen sleep problems with habits that promote sound sleep. There will be 6 intervention sessions over an 8-week period. The first two sessions are consecutive weekly in-person sessions followed by a rest week. The third session is conducted remotely by phone, followed by another rest week. The three remaining sessions are weekly and conducted remotely.
  Arms: CBT-I + BWL
Behavioral: Sleep Education — EDU involves learning behavioral treatment information about sleep that is widely available to patients and practitioners. The program will parallel the CBT-I intervention in schedule, number, and length of sessions.
  Arms: EDU + BWL

SUMMARY:
This is a randomized pilot study to better understand the relationships among insomnia, weight loss, and breast cancer. This study will assess the effectiveness of a sleep intervention prior to a web- and phone-based weight loss program.

DETAILED DESCRIPTION:
Participants are women with a diagnosis of early stage breast cancer (ESBC), a BMI ≥25, and insomnia. A total of 30 participants will be randomized to either cognitive behavioral therapy for insomnia and behavioral weight loss (CBT-I+BWL) or a sleep education program and behavioral weight loss (EDU+BWL). Measures will be collected at baseline, 8 weeks (after the CBT-I or EDU program) and at 3 and 6 months after starting BWL. The primary outcome will be % total weight loss. Additionally, eating behaviors, physical activity, and sleep parameters will be carefully assessed.

The sleep intervention phase of the study includes 6 sessions over 8 weeks (2 in-person, followed by 4 phone or videoconferencing sessions), and the BWL intervention includes 15 sessions over 6 months (1 in-person, 14 by phone or videoconference). Participants will be given physical activity trackers and will use a dietary app to record their food intake. There are 4 in-person assessment visits (baseline/randomization, 8-week follow up, 3-month follow up, 6-month follow up). These assessment visits are coordinated with in-person sleep and weight loss intervention visits. Some of the measures that will be recorded throughout the study include: height, weight, anthropometric measures (waist/hip measurements), sleep diaries, and self-report measures.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years of age or older
* Histologically-confirmed ductal carcinoma in-situ (DCIS) or stage I-III invasive carcinoma of the breast
* Current BMI ≥ 25 kg/m2 and weight ≤ 400 lbs
* Willing to lose 10% of body weight
* Diagnosed with current breast cancer >3 and <60 months from planned baseline visit date
* Completed local therapy (i.e. surgery and radiation therapy) and any planned preoperative or adjuvant chemotherapy within >3 prior to enrollment
* Diagnosed with insomnia or reports sleep problems
* Has daily access to the internet and/or smartphone

Exclusion Criteria:

* Serious/uncontrolled condition likely to hinder accurate measurement of weight or sleep, such as bipolar I, seizure disorders, autoimmune disease, etc., or a medical condition that makes physical activity unsafe
* Current use of weight loss medications or sleeping aids
* Current enrollment in a sleep or weight loss program
* Sleep disorder other than insomnia
* Plan to become pregnant within next 12 months, or lactating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Percent Weight loss | Change from Baseline, 8 weeks, 3 months and 6 months
  The primary outcome will be percent (%) weight loss. All subjects who are randomized will be included in the analysis of the primary outcome. Weight will be measured according to standardized BMI and anthropometric procedures (hip/waist ratio). For the primary aim, comparing the effects of CBT-I+BWL and EDU+BWL on % weight loss at 3 and 6 months, we will model outcomes (at 3 months & 6 mos.) as a function of baseline level, treatment assignment, time, and their interaction. The interaction term represents the between-group difference in change over time on the outcome.

SECONDARY OUTCOMES:
Sleep continuity as measured by wake after sleep onset (WASO) | Change from Baseline, 8 weeks, 3 months and 6 months
  WASO will be measured in minutes. Sleep continuity will be measured using actigraphs and sleep diaries at baseline, 8 weeks, 3 months, and 6 months. For this aim, evaluating the extent to which short-term sleep continuity improvements (8 wk and 3 mo) are associated with improvements in daily physical activity and dietary quality/quantity and determining their association with 3- and 6-month weight changes, we will model between-group differences in the short-term trajectory of change for the primary sleep continuity measures, actigraphy TST and WASO.
Sleep continuity as measured by total sleep time (TST) | Change from Baseline, 8 weeks, 3 months and 6 months
  TST will be measured in minutes. Sleep continuity will be measured using actigraphs and sleep diaries at baseline, 8 weeks, 3 months, and 6 months. For this aim, evaluating the extent to which short-term sleep continuity improvements (8 wk and 3 mo) are associated with improvements in daily physical activity and dietary quality/quantity and determining their association with 3- and 6-month weight changes, we will model between-group differences in the short-term trajectory of change for the primary sleep continuity measures, actigraphy TST and WASO.
Sleep continuity as measured by sleep efficiency (SE) | Change from Baseline, 8 weeks, 3 months and 6 months
  Sleep efficiency is measured as the ratio of total sleep time (TST) compared to the total time spent in bed (TST / time in bed). This is measured in percent of total time spent in bed, asleep.
  Sleep continuity will be measured using actigraphs and sleep diaries at baseline, 8 weeks, 3 months, and 6 months.
Sleep continuity as measured by sleep latency (SL) | Change from Baseline, 8 weeks, 3 months and 6 months
  Sleep latency is the time it takes to transition from full wakefulness to sleep. This is measured in minutes. Sleep continuity will be measured using actigraphs and sleep diaries at baseline, 8 weeks, 3 months, and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Janelle Coughlin, Ph.D., Principal Investigator — Associate Professor
Locations (1):
- Johns Hopkins University, Bayview Medical Campus, Baltimore, Maryland, United States